CLINICAL TRIAL: NCT05199324
Title: Early Oral Step-down Antibiotic Therapy Versus Continuing Intravenous Therapy for Uncomplicated Gram-negative Bacteraemia (the INVEST Trial)
Brief Title: Early Oral Step-down Antibiotic Therapy for Uncomplicated Gram-negative Bacteraemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Singapore Clinical Research Institute, Singapore (Unknown); National University Hospital, Singapore (Other); Singapore General Hospital (Other); Changi General Hospital (Other); Ng Teng Fong General Hospital, Singapore (Unknown); Sengkang General Hospital, Singapore (Unknown); Royal Brisbane and Women's Hospital, Australia (Unknown); Royal Melbourne Hospital, Australia (Unknown); University Malaya Medical Centre, Malaysia (Unknown); Samsung Medical Center, South Korea (Unknown); Princess Alexandra Hospital, Australia (Unknown); Gold Coast University Hospital, Australia (Unknown); Ampang Hospital, Malaysia (Unknown); Sungai Buloh Hospital, Malaysia (Unknown); Universiti Kebangsaan Medical Centre, Malaysia (Unknown); Istanbul Medipol University Hospital (Other); Rambam Hospital, Israel (Unknown); Sheba Medical Centre, Israel (Unknown); IRCCS Policlinico di Sant'Orsola, University Alma Mater Studiorum of Bologna, Italy (Unknown); Monaldi Hospital, Italy (Unknown); University Hospital of Pisa, Italy (Unknown); IRCCS San Raffaele (Other); University General Hospital of Patras, Greece (Unknown); Hospital del Mar, Parc de Salut MAR, Spain (Unknown); American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSRB 2021/00764
Record Dates: First submitted 2021-12-21; First posted 2022-01-20 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Gram-negative Bacteraemia
Keywords: Gram-negative bacteraemia; Early stepdown to oral antibiotics; Oral fluoroquinolones; Oral trimethoprim-sulfamethoxazole; Continuing intravenous antibiotics; Health economic evaluation
MeSH Terms: interventions — Fluoroquinolones; Ciprofloxacin; Trimethoprim, Sulfamethoxazole Drug Combination; Cefazolin; Ceftriaxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early step-down to oral antibiotic therapy (Experimental): The oral antibiotic options are fluoroquinolones (most commonly, ciprofloxacin) or trimethoprim-sulfamethoxazole. The recommended doses for patients with normal renal function would be ciprofloxacin 750 mg twice daily (if body weight ≥70 kg) or ciprofloxacin 500 mg twice daily (if body weight <70 kg) or trimethoprim-sulfamethoxazole 5 mg/kg (for trimethoprim component) every 12 hourly or trimethoprim-sulfamethoxazole (160 mg / 800 mg; double strength) two tablets twice daily. Doses may be adjusted in the setting of renal dysfunction. The recommended treatment duration by the study team is 7 days of active antibiotics (including empiric therapy), although treatment regimen may be longer than 7 days due to regimen extension or requirement for prolonged regimen as clinically indicated.
  Interventions: Drug: Oral fluoroquinolones (most commonly, ciprofloxacin) or oral trimethoprim-sulfamethoxazole
- Continuing intravenous antibiotic therapy (Active Comparator): The intravenous antibiotic(s) to be administered will be determined by the treating doctor according to what would be considered standard of care in the hospital site. Commonly used intravenous antibiotics (and doses) for treatment of Gram-negative bacteraemia include ceftriaxone 2 g daily or cefazolin 2 g three times daily. The recommended treatment duration by the study team is 7 days of active antibiotics (including empiric therapy), although treatment regimen may be longer than 7 days due to regimen extension or requirement for prolonged regimen as clinically indicated.
  Interventions: Drug: Standard of care intravenous antibiotics (e.g. ceftriaxone, cefazolin)

INTERVENTIONS:
Drug: Oral fluoroquinolones (most commonly, ciprofloxacin) or oral trimethoprim-sulfamethoxazole — Clinically stable / non-critically ill inpatients with uncomplicated Gram-negative bacteraemia randomised to the intervention arm will be switched early to oral antibiotics (within 72 hours from index blood culture collection)
  Other Names: Fluoroquinolones (most commonly, cipro); Bactrim
  Arms: Early step-down to oral antibiotic therapy
Drug: Standard of care intravenous antibiotics (e.g. ceftriaxone, cefazolin) — Clinically stable / non-critically ill inpatients with uncomplicated Gram-negative bacteraemia randomised to the standard arm will continue to receive an active intravenous antibiotic therapy for at least another 24 hours post-randomisation before clinical re-assessment and decision making by the treating doctor
  Other Names: Rocephin; Kefzol
  Arms: Continuing intravenous antibiotic therapy

SUMMARY:
Current management of uncomplicated Gram-negative bacteraemia entails prolong intravenous (IV) antibiotic therapy with limited evidence to guide oral conversion. This trial aim to evaluate the clinical efficacy and economic impact of early step-down to oral antibiotics (within 72 hours from index blood culture collection) versus continuing standard of care IV therapy (for at least another 24 hours post-randomisation) for clinically stable / non-critically ill inpatients with uncomplicated Gram-negative bacteraemia.

DETAILED DESCRIPTION:
This is an international, multicentre, randomised controlled, open-label, phase IV, non-inferiority trial with a non-inferiority margin of 6%. Eligible participants must be clinically stable / non-critically ill inpatients over the age of 18 years old (in Singapore, 21 years and above) with uncomplicated Gram-negative bacteraemia. Randomisation into the intervention or standard arms will be performed with 1:1 allocation ratio according to a randomisation list prepared in advance using a secure online randomisation system. Randomisation will be stratified by country and random sequence will be generated using random permuted blocks of unequal length. Participants randomised to the intervention arm (within 72 hours from index blood culture collection) will be immediately converted to oral fluoroquinolones (most commonly, ciprofloxacin) or oral trimethoprim-sulfamethoxazole. In the event of microbiological or clinical failure of the oral antibiotic treatment, escalation to IV antibiotics may be initiated at any time point post-randomisation. Participants randomised to the standard arm should continue to receive an active IV therapy for at least another 24 hours post-randomisation before clinical re-assessment and decision making by the treating doctor. All the study drugs (and dosage) would be routinely used in clinical practice and will be ordered/dispensed from the hospital pharmacy as per site institutional practice. The recommended treatment duration by the study team is 7 days of active antibiotics (including empiric therapy), although treatment regimen may be longer than 7 days if clinically indicated. Participants may be discharged home or to OPAT at any time post-randomisation.

ELIGIBILITY:
Inclusion Criteria:

1. One or more set(s) of blood cultures positive for Gram-negative bacteria (GNB) associated with evidence of infection
2. Able to be randomised within 72 hours of index blood culture collection
3. Age ≥18 years (≥21 in Singapore)
4. Latest Pitt bacteraemia score <4
5. Patient or legal representative is able to provide informed consent

Exclusion Criteria:

1. Established uncontrolled focus of infection, including but not limited to:

   * Undrained abdominal abscess, deep seated intra-abdominal infection and other unresolved abdominal sources requiring surgical intervention
   * Central nervous system abscess (patients with focal neurology should have cranial CT prior to enrolment)
   * Undrained moderate-to-severe hydronephrosis
2. Complicated infections, including but not limited to:

   * Necrotising fasciitis
   * Empyema
   * Central nervous system infections and meningitis
   * Endocarditis / endovascular infections
3. Septic shock as defined by systolic blood pressure <90 or mean arterial pressure <70 mmHg despite adequate fluid resuscitation or need for inotropic/vasopressor support
4. Polymicrobial bacteraemia involving Gram-positive pathogens or anaerobes (defined as either growth of 2 or more different microorganism species in the same blood culture, or growth of different species in 2 or more separate blood cultures within the same episode [<48 hours] and with clinical or microbiological evidence of the same source)
5. Bacteraemia is due to a vascular catheter or intravascular materials (e.g. pacing wire, vascular graft) that cannot be removed
6. Specific Gram-negative pathogens that cannot be effectively treated with fluoroquinolones or trimethoprim-sulfamethoxazole, including but not limited to, Burkholderia spp. and Brucella spp.
7. Index GNB with resistance to fluoroquinolones AND trimethoprim-sulfamethoxazole
8. Hypersensitivity to fluoroquinolones AND sulphur drugs as defined by history of rash, urticaria, angioedema, bronchospasm, circulatory collapse or significant adverse reaction following prior administration
9. Unable to consume or absorb oral medications for any reason or unsuitable for ongoing IV therapy (e.g. no intravenous access)
10. Severely immunocompromised in the opinion of the treating doctor, including but not limited to, medical conditions such as:

    * Active leukaemia or lymphoma
    * Aplastic anaemia
    * Bone marrow transplant within two years of transplantation or transplants of longer duration still on immunosuppressive drugs or with graft-versus-host disease
    * Congenital immunodeficiency
    * HIV/AIDS with CD4 lymphocyte count <200
    * Neutropenia or expected post-chemotherapy neutropenia within 14 days from the time of screening, defined as absolute neutrophil count < 500 cells/μL
11. Women who are known to be pregnant or breast-feeding
12. Treatment is not with intent to cure the infection (i.e. palliative care)
13. Unable to collect patient's follow-up data for at least 30 days post-randomisation for any reason
14. Treating doctor deems enrolment into the trial is not in the best interest of the patient
15. Previous enrolment in this trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  All-cause mortality at day 30 post-randomisation

SECONDARY OUTCOMES:
14-day and 90-day mortality | 90 days
  All-cause mortality at days 14 and 90 from the time of randomisation
Duration of survival by day 90 | 90 days
  Duration of survival (in days) from the time of randomisation until day 90
Number of days on IV antibiotic therapy in the total index hospitalisation | 90 days
  Number of days on IV antibiotic therapy in the total index hospitalisation (including outpatient parenteral antibiotic therapy [OPAT]) for surviving participants from the time of randomisation until i. hospital discharge and ii. day 90
Number of days alive and free of antibiotics by day 90 | 90 days
  Number of days alive and free of antibiotics (i. for all antibiotics and ii. for IV antibiotics) between the time of randomisation and day 90
Adverse events from the time of randomisation until day 90 | 90 days
  Solicited adverse events include Clostridioides difficile-associated diarrhoea, peripherally inserted central catheter and other central venous catheter complications (such as catheter-related bloodstream infection, catheter-related superficial or deep venous thrombosis/thrombophlebitis, catheter blockage, and exit site infection) requiring line removal during index hospitalisation (including OPAT) from the time of randomisation, and liver function test abnormalities or acute kidney injury
Change in treatment strategy between the time of randomisation and day 30 | 30 days
  Change in treatment strategy (e.g. switch to IV antibiotics from allocated oral antibiotics or vice versa) between the time of randomisation and day 30 due to: (i) an adverse event deemed by the treating doctor to be of sufficient severity to change treatment strategy, or (ii) presumed lack of efficacy of treatment strategy according to the judgement of treating doctor
Time to being discharged alive from the total index hospitalisation between the time of randomisation and day 90 | 90 days
  Time to being discharged alive from the total index hospitalisation (including OPAT and hospital in the home) between the time of randomisation and day 90 (note: any death occurrence within 90 days will be considered '90 days')
Number of days alive and not in hospital by day 90 | 90 days
  Number of days alive and not in hospital (including OPAT) between the time of randomisation and day 90
Readmission or extended hospitalisation by day 90. | 90 days
  Readmission is defined as a new hospitalisation for any cause occurring after discharge from the index hospitalisation. Extended hospitalisation is defined as >14 days of hospital LOS starting from the day of randomisation.
Health economic evaluation | 90 days
  Health economic evaluation includes calculation of estimated total healthcare cost (from healthcare system and patient perspective) by day 90
Assessment of patient's quality of life | 90 days
  Assessment of patient's quality of life via EQ-5D-5L on screening day, end of treatment day, and day 90

CONTACTS AND LOCATIONS:
Overall Officials: David Lye, MBBS, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee IR, Tong SYC, Davis JS, Paterson DL, Syed-Omar SF, Peck KR, Chung DR, Cooke GS, Libau EA, Rahman SBA, Gandhi MP, Shi L, Zheng S, Chaung J, Tan SY, Kalimuddin S, Archuleta S, Lye DC. Early oral stepdown antibiotic therapy versus continuing intravenous therapy for uncomplicated Gram-negative bacteraemia (the INVEST trial): study protocol for a multicentre, randomised controlled, open-label, phase III, non-inferiority trial. Trials. 2022 Jul 19;23(1):572. doi: 10.1186/s13063-022-06495-3. PMID 35854360